CLINICAL TRIAL: NCT03821337
Title: An Exploratory Investigation Utilizing Repetitive Transcranial Magnetic Stimulation (rTMS) as a Tool to Decrease Pain and Improve Functioning in Veterans With Opioid Use Disorder
Brief Title: Transcranial Magnetic Stimulation (rTMS) as a Tool to Decrease Pain and Improve Functioning
Acronym: TMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 placed all Charleston VA projects on hold. Recently gained approval to open studies with COVID-19 precautions
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3006-P; RX003006 (Other Grant/Funding Number: Department of Veterans Affairs); Pro00084970 (Other: MUSC IRB)
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Opioid Use Disorder
Keywords: Opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Double-blind, Randomized, Placebo-Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rTMS (Experimental): Participants will receive 18 sessions of active rTMS delivered at 120% rMT.
  Interventions: Device: repetitive Trans Magnetic Stimulation
- Sham TMS (Placebo Comparator): Participants will receive 18 sessions of sham rTMS delivered through an inactive coil.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: repetitive Trans Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that is able to alter cortical excitability and is FDA-approved to treat Major Depressive Disorder. Magnetic fields pass unimpeded through the scalp, skull and meninges, and can directly excite cortical areas.
  Other Names: rTMS
  Arms: rTMS
Device: Sham TMS — Sham sessions will be delivered using an electronic sham system consisting of a coil that mimics the appearance and sound of TMS, combined with a TENS device which produces a small electric shock mimicking the feeling of real rTMS. This type of sham has been demonstrated to be indistinguishable from real rTMS, has been well tolerated (George et al., 2010; George et al., 2014) and successfully used in other clinical trials (Borckardt et al., 2008; Arana et al., 2008). During each session of rTMS the investigators will present a series of opioid related images, including those utilized in previous studies (Garland et al., 2015; Garland & Howard, 2014).
  Arms: Sham TMS

SUMMARY:
Despite the availability of opioid replacement therapies, many opioid use disordered Veterans are not able to remain abstinent. Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive neuromodulation technique with a consistent, rapidly expanding literature base reporting positive outcomes in substance using populations. This pilot application will investigate a novel multi-session rTMS paradigm to determine feasibility and tolerability of this intervention in opioid use disordered Veterans.

DETAILED DESCRIPTION:
Opioid use disorders (OUDs) are common among Veterans. Despite the availability of opioid replacement therapies, many individuals continue to abuse opioids and relapse rates remain high. Veterans are nearly twice as likely to die from accidental opioid overdose than the general population. Approximately 60% of Veterans returning from the Middle East and more than 50% of older Veterans in the VA health care system have chronic pain. Further, post-traumatic stress disorder, a common comorbidity in the Veteran population, has been shown to negatively impact early engagement and retention of individuals in OUD treatment. As is the case with other substance use disorders, opioid craving is commonly described by abstinent patients whether or not they are stabilized on buprenorphine. Subsequently, a treatment that reduces pain and craving, while also improving early engagement and retention in treatment, would improve recovery from opioid addiction. Repetitive Transcranial Magnetic Stimulation (rTMS) is capable of non-invasively altering cortical function. rTMS is an FDA-approved treatment for major depressive disorder. Preliminary evidence suggests that rTMS can also reduce pain in chronic pain conditions and craving in substance use disorders. Single sessions of rTMS produce small temporary effects, while multiple sessions of rTMS result in larger, more durable effects. The investigators' group recently completed a blinded, sham-controlled crossover trial in non-treatment seeking OUD participants. A single session of rTMS reduced cue-induced craving and increased thermal pain thresholds. Given that multiple sessions of rTMS produce larger and more durable treatment effects than single sessions of rTMS, it follows that multiple treatment sessions applied to OUD patients may result in a clinically relevant reduction in pain and cue-induced craving, which could improve clinical and functional outcomes.

In this SPiRE pilot proposal, the investigators will perform a randomized, double-blind, sham-controlled trial delivering an accelerated course of rTMS to a cohort of OUD Veterans with chronic pain receiving treatment through the Ralph H. Johnson VA Medical Center Substance Treatment and Recovery program. The goal of this proposal is to evaluate the feasibility and acceptability of delivering rTMS to the dorsolateral pre-frontal cortex in Veterans with OUD and chronic pain. The investigators will also preliminarily explore the feasibility of evaluating potential outcome measurements in preparation for a larger trial, including abstinence, treatment retention, community reintegration and functional outcomes, pain, and opioid craving. Positive results from this pilot project will inform a future MERIT application and have the potential to significantly improve treatment outcomes in this difficult to treat Veteran population.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Participants must meet moderate to severe DSM-5 criteria for OUD. While individuals may also meet criteria for use disorders of other substances (with the exception of alcohol or benzodiazepines), they must identify opioids as their primary substance of abuse.
* Participants must report chronic pain for at least the past three months and have a Brief Pain Inventory score.
* Participants must be receiving treatment through the STAR program.

Exclusion Criteria:

* Participants who are pregnant.
* Participants with a history of/or current psychotic disorder.
* Participants with a history of dementia or other cognitive impairment.
* Participants with active suicidal ideation, or a suicide attempt within the past 90 days will be excluded.
* Participants with contraindications to receiving rTMS (including a history of seizures, or any implanted metal above the neck).
* Those with unstable general medical conditions.
* Those who are currently using naltrexone or tramadol.
* Those with current alcohol or benzodiazepine use disorders due to increased risk of seizure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee L. Mcrae-Clark, PharmD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rTMS | Sham TMS
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Veterans being treated for opioid use disorder. Only one subject completed rTMS sessions and they were in the rTMS group.
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS | Sham TMS | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55 (NA) — Standard Deviation is not calculable for 1 participant. |  | 55 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Retention: Total Number of rTMS Sessions Completed
Description: Total number of rTMS sessions completed out of 6 sessions per day for three days over a three week period.
Time Frame: Through study completion, an average of 3 weeks
Population: Veterans being treated for opioid use disorder. Only one subject completed rTMS sessions and they were in the active rTMS group.
Measure: Number; unit: Sessions completed
Arm/Group | rTMS | Sham TMS
Number analyzed (Participants) | 1 | 0
Sessions completed | 18 |

2. Primary Outcome: Tolerability: The Total Number of Treatment Emergent Adverse Events
Description: Number of adverse events experienced by Veterans receiving medication assisted treatment for opioid use disorder who undergo 18 sessions of active or sham rTMS.
Time Frame: Through study completion, an average of 3 weeks
Population: Veterans receiving medication assisted treatment for opioid use disorder.
Measure: Number; unit: Adverse Events
Arm/Group | rTMS | Sham TMS
Number analyzed (Participants) | 1 | 0
Adverse Events | 1 |

ADVERSE EVENTS:
Time Frame: Three weeks of once weekly treatment sessions.
Description: 0 participants were at risk for adverse events in the sham condition because no participants were randomized to that condition.
Arm/Group | rTMS | Sham TMS
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=1) | Sham TMS (N=0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03821337/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03821337/ICF_001.pdf